CLINICAL TRIAL: NCT06267261
Title: Clinical Evaluation of Surgical Face Mask Efficacy in Reducing Asthma and Rhinitis Symptoms in Birch-allergic Subjects in ALYATEC Environmental Exposure Chamber
Brief Title: Efficacy of Face Mask in Reducing Respiratory Allergic Symptoms in Birch-allergic Subjects in ALYATEC Exposure Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyatec (Industry)
Collaborators: Medicom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KOL-001
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Allergic Asthma; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with face mask (Experimental): Birch pollen allergen exposure in ALYATEC chamber with face mask
  Interventions: Device: KOLMI® surgical face mask (OP-Air)
- Patients without face mask (No Intervention): Birch pollen allergen exposure in ALYATEC chamber without face mask

INTERVENTIONS:
Device: KOLMI® surgical face mask (OP-Air) — 12 subjects are exposed to birch pollen allergen in ALYATEC EEC while wearing a KOLMI® surgical face mask (OP-Air)
  Arms: Patients with face mask

SUMMARY:
There is no clinical evidence that face masks are efficient in birch pollen-induced asthma. As the use of face masks has become widespread worldwide to limit the spread of SARS-CoV-2, this study aims to demonstrate the clinical efficacy of medical masks in patients allergic to birch in the same way that clinical trial with drugs.

DETAILED DESCRIPTION:
All patients should have positive skin prick tests and specific IgE to birch at screening visit. 24 patients with asthma response during 1-hour baseline exposure to airborne Bet v 1 in ALYATEC environmental exposure chamber.will be randomized into 2 groups: with (n=12) and without (n=12) a KOLMI® surgical face mask (OP-Air), for a 6-hour exposure to birch allergen.

Allergic symptoms will be observed during the 6-hour exposure and compared between the 2 different groups (with and without face mask) to evaluate the efficacy of the face mask.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects who signed the written informed consent,
* Subjects covered by health social identification number,
* Subjects able to understand and complete study-related procedures,
* Subjects reported history of symptomatic birch pollen allergen-triggered asthma (GINA1) with associated allergic rhinitis,
* Positive skin prick test (SPT) with cat hair extract with mean wheal diameter ≥ 5 mm compared to negative control (NaCl reaction < 2 mm),
* Positive sIgE tests for birch tree pollen and Bet v 1 (≥0.7 kUa/L),
* Subjects with FEV1 ≥ 70% predicted at screening and before allergen exposure,
* Subjects with at least one drop in FEV1 ≥20% during the 1-hour baseline exposure
* ACT≥ 20,
* Women of childbearing potential with a negative pregnancy test throughout the study period and a highly effective contraception: oral contraceptives, condom with spermicide, intrauterine device, bilateral tubal ligation, vasectomized partner.

Main Exclusion Criteria:

* Allergen immunotherapy to birch pollen allergen for more than 1 month in the 3 years prior to the screening visit,
* Ongoing allergen immunotherapy to another allergen,
* History of anaphylactic reactions to birch allergen exposure or birch allergen immunotherapy,
* History of anaphylactic reactions to another allergen in the last 6 weeks before inclusion,
* Nasal polyposis, deviation of nasal septum or diagnosis of uncontrolled non-allergic rhinitis,
* Subjects allergic to indoor environmental allergens (molds, house dust mite allergens) with obvious exposure to these allergens causing allergic symptoms,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Time to early asthma response (EAR) | 0 to 6 hours
  The efficacy of face mask is evaluated by the time necessary to observe an EAR during birch pollen allergen exposure in EEC

SECONDARY OUTCOMES:
Frequency of EAR and late asthma response (LAR) | 0 to 6 hours (EAR) - 3 to 24 hours after exposure (LAR)
  The efficacy of face mask is evaluaed by the frequency of EAR and LAR during and after birch pollen allergen exposure in EEC
Severity of EAR and LAR | 0 to 6 hours (EAR) - 3 to 24 hours after exposure (LAR)
  The efficacy of face mask is evaluated by the maximum percentage of drop of FEV1during and after EEC exposure
Nasal Symptoms | 0 to 6 hours. (Total Nasal Symptoms Score from 0 to 12, 0 being the worse and 12 the better score)
  The efficacy of face mask is evaluated with specific questionnaire (Total Nasal Symptoms Score - TNSS)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric de Blay, Pr, Principal Investigator — Chest Diseases Department, Strasbourg University Hospital, France
Locations (1):
- ALYATEC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study results — https://www.em-consulte.com/article/1557183/evaluation-clinique-de-l-efficacite-d-un-masque-ch